CLINICAL TRIAL: NCT03514134
Title: Modifying (Phase I) and Evaluating (Phase II) Virtual Reality Job Interview Training for Youth in Transition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Wisconsin, Madison (Other); SIMmersion, LLC (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Matthew Smith, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00129575; 5R34MH111531-03 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-05-02 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Services as usual + Virtual Reality Job Interview Training (Experimental): In addition to the services as usual comparator, participants will participate in Virtual Reality Job Interview Training.
  Interventions: Behavioral: Virtual Reality Job Interview Training; Behavioral: Services as Usual
- Services as Usual (Active Comparator): Study participants will be receiving their community-based or school-based services as usual that may include but is not limited to vocational skill training, daily living skill training, and social skill training.
  Interventions: Behavioral: Services as Usual

INTERVENTIONS:
Behavioral: Virtual Reality Job Interview Training — Students will engage in didactic training related to strategies to perform well during a job interview as well as repeated practice with a virtual hiring manager. Throughout and after completion of the virtual interviews, participants will receive feedback on their performance.
  Arms: Services as usual + Virtual Reality Job Interview Training
Behavioral: Services as Usual — Study participants will be receiving their community-based or school-based services as usual that may include but is not limited to vocational skill training, daily living skill training, and social skill training.

SUMMARY:
The unemployment rate is quite high among adults with an autism spectrum disorder (ASD). Inadequate transition planning during high school and gaps between vocational needs and availability of evidence-based services help explain the struggles of transition-age youth at obtaining employment. There is a paucity of research on developing and evaluating services to support the transition to the work force after graduating from high school. The lack of available resources to support transition-age youth with an ASD speaks to the need to develop interventions that ameliorate obstacles to employment and help support the transition to the work force. Due to the social deficits characterizing ASD innovative interventions could target preparing job interview skills for students facing the transition to employment as the job interview is a critical gateway to securing a job offer. Thus, the overarching goal of this study is to modify an existing virtual reality job interview skills training program for use in high school students with ASD and to test the feasibility and effectiveness of conducting this intervention in a high school setting via a small controlled trial. Thus, study's first aim is to modify the existing 'Virtual Reality Job Interview Training' program to meet the specific needs of high school seniors with ASD. This will accomplish this by conducting in depth interviews with high school students with ASD and their vocational counselors to solicit feedback to modify the current training's learning goals, content, usability, and simulated interview scripts to meet the specific needs of transition age youth. An expert panel will determine the final modifications to the training program based on the results of the qualitative data analysis and their own views of the program. Second aim of the study is to conduct a pilot trial to evaluate the feasibility, acceptability, portability, fidelity and preliminary effectiveness of the modified intervention in a randomized controlled trial. This study will also explore potential mechanisms for effectiveness and collect pilot implementation data.

ELIGIBILITY:
Inclusion Criteria:

1. 16-26 years old and enrolled in high school or post-high school transition programming;
2. Educational Diagnosis of autism spectrum disorder using the Social Responsivity Scale 2nd Edition28, or a diagnosis of cognitive impairment, emotional disability, educational impairment or other health impairment according to the students Individualized Education Plan (IEP). They may have diagnosis of autism spectrum disorder as indicated in their IEP/school plan, or as indicated by a parent;
3. Fluency in English with at least a 3rd grade reading level (confirmed with the Wide Range Achievement Test);
4. Currently receiving transitional services as specified in IEP or other;
5. Willing to be video-recorded; and
6. Willing and able to provide informed consent.

Exclusion Criteria:

1. Has an uncorrected hearing or visual problem that prevents him or her from using the training.
2. Has a medical illness that compromises their cognition (for example, moderate to severe traumatic brain injury)

Inclusion and exclusion criteria is subject to PI discretion. Some students may still be enrolled after discussion with the teacher if it is determined that they still might be able to participate despite matching exclusion criteria, or not meeting all of the inclusion criteria. These cases will be documented and reported to IRB.

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smith, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
Started | 23 | 48
Completed | 23 | 47
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training | Total
Number analyzed (Participants) | 23 | 48 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.4 (2.6) | 19.8 (3.0) | 19.7 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 20 | 38 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 13 | 26 | 39
  Black/African American | 8 | 11 | 19
  Latinx | 0 | 6 | 6
  More than one race | 2 | 2 | 4
  Asian American | 0 | 2 | 2
  Native American | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 48 | 71
Social Responsiveness Scale (Second Edition) [Mean (Standard Deviation); unit: T-Score] — Measure was collected by parents/teachers about the autism participants. These are the total T-Scores indicating deficiencies in reciprocal social behavior. The T-Score has a mean of 50 points with a standard deviation of 10 points. Greater than or equal to 76T means that deficiencies in reciprocal social behavior are clinically significant and strongly associated with a clinical diagnosis of autism. Ranges 66T-75T indicate Moderate deficiencies, 60T-65T indicate Mild deficiencies, and 59T or lower indicate Normal. There were 65 questions on a scale from 1 (not true) to 4 (almost always true).
  T-Score | 63.9 (14.1) | 65.7 (13.2) | 65.2 (13.4)
Current grade [Count of Participants; unit: Participants]
  Sophomore | 2 | 3 | 5
  Junior | 3 | 6 | 9
  Senior | 6 | 14 | 20
  Transitional year | 12 | 25 | 37
Co-occuring IDEA categorizations [Count of Participants; unit: Participants]
  Other health impairment | 5 | 10 | 15
  Specific learning disability | 3 | 5 | 8
  Cognitive impairment | 2 | 9 | 11
  Emotional disturbance | 3 | 5 | 8
Cognitive ability [Mean (Standard Deviation); unit: T-Score] — Cognitive ability was measured using the National Institute of Health (NIH) Toolbox. The Fluid Composite score was created by averaging the standard scores of 5 of the subtests, then deriving standard scores based on the new distribution. Crystallized Composite Score was created by using 2 subtests, with the score being created by averaging the standard scores of each of the measures, and then deriving standard scores based on the new distribution. Higher scores indicate higher levels of functioning for both composites. These are T-Score averages, with a normative mean of 50 and SD of 10.
  T-Score
    Fluid Cognition Composite | 33.3 (13.1) | 29.6 (10.9) | 30.8 (11.7)
    Crystalized Cognition Composite | 40.1 (11.5) | 42.7 (12.4) | 41.9 (12.1)
Vocational history [Count of Participants; unit: Participants]
  Ever had a job interview | 8 | 14 | 22
  Ever employed at competitive, integrated job | 5 | 16 | 21
  Currently employed at competitive, integrated job | 1 | 5 | 6
Mood and Feelings Questionnaire [Mean (Standard Deviation); unit: units on a scale] — This survey measures depressive symptoms and was 13 items with higher scores indicating higher depressive symptoms. Items were rated on a scale of 0 (Not True), 1 (Sometimes), or 2 (True). The range of scores was 0-26.
  units on a scale | 4.7 (4.1) | 5.7 (4.1) | 5.4 (4.1)
Adult and Child Behavior Checklist [Mean (Standard Deviation); unit: T-Score] — Internalizing and externalizing behaviors were measured with the standardized child behavior checklist (CBCL) and adult behavior checklist (ABCL). These forms rated 118 trait behaviors reflecting internalizing behaviors (anxious/depressed, somatic complaints, withdrawn, etc.) and externalizing behaviors (rule-breaking, aggressive behavior, etc.). Behaviors were rated on a three-point scale of 0 (not true) to 1 (very true), where higher total t-scores reflected more behaviors. Internalizing and Externalizing t-scores both have a mean of 50 and a standard deviation of 10.
  T-Score
    Internalizing Behaviors | 54.9 (10.1) | 59.5 (10.3) | 58.0 (10.3)
    Externalizing Behaviors | 51.6 (11.1) | 52.0 (10.3) | 51.9 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Job Interview Skills
Description: Interviewing skills will be measured using a role-play measure in which subjects act out one job interview scenario with trained actors. Interviews will be video recorded and scored. There is one mock interview and pre-test and one mock interview at post-test. The method of assessment is the job interview skills rating scale as measured by the Mock Interview Rating Scale, which has 14 items with each item ranging from 1 (Unlikely) to 7 (Very Likely). Possible scores range from 14 to 98, with higher scores indicating better interview skills.
Time Frame: Collected at Pre-Test and Post-Test visits (within approximately 1 month of active treatment)
Population: Performance on 2 Mock Job Interviews collected at pre-test and post-test
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
Number analyzed (Participants) | 23 | 48
score on a scale
  Pre-test | 45.9 (1.9) | 46.8 (1.3)
  Post-test | 43.6 (1.9) | 49.6 (1.3)
Statistical Analysis 1: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; Test type: Superiority; p < 0.001, ANCOVA; Repeated measures ANCOVA

2. Secondary Outcome: Job Interview Self-Efficacy
Description: 9 item self-report consisting of 11 items on a 5-point Likert-type scale, with 1 indicating "Not at all" and 5 indicating "Very True". The range of scores is from 11 to 55, with higher scores indicating more self-efficacy/motivation to complete job interviews, which is a better outcome.
Time Frame: Collected at Pre-Test and Post-Test visits (within approximately 1 month of active treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
Number analyzed (Participants) | 23 | 48
score on a scale
  Pre-test | 45.9 (3.4) | 47.2 (2.6)
  Post-test | 44.3 (3.1) | 43.5 (2.4)
Statistical Analysis 1: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; Test type: Superiority; p = 0.358, ANCOVA; Repeated measures ANCOVA

3. Secondary Outcome: Change in Job Interview Anxiety
Description: 15 item self-report using a modified version of the brief Personal Report of Public Speaking Apprehension (PRSPA; McCroskey, 1970). After reviewing the brief PRSPA, we selected and reframed 10 items using a three point Likert-type scale (0 = "not at all," 1 = "sometimes," and 2 = "often"). Higher scores indicated higher anxiety, and scores could range from 0 to 26.
Time Frame: Collected at Pre-Test and Post-Test visits (within approximately 1 month of active treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
Number analyzed (Participants) | 23 | 48
score on a scale
  Pre-test | 5.0 (4.7) | 7.0 (4.1)
  Post-test | 4.4 (4.4) | 5.7 (3.8)
Statistical Analysis 1: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; Test type: Superiority; p = 0.029, ANCOVA; Repeated measures ANCOVA

4. Secondary Outcome: Competitive Employment
Description: Obtained a part-time or full-time community-based job as completed via a self-report measure yes/no question. This survey could have been completed by either participants themselves, parents, or teachers.
Time Frame: Collected at pre-test and at 6 months after completing Post-Test Visit
Population: Competitive Employment
Measure: Count of Participants; unit: Participants
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
Number analyzed (Participants) | 23 | 48
Participants | 0 | 12
Statistical Analysis 1: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; Test type: Superiority; p < 0.01, Chi-squared
Statistical Analysis 2: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; Test type: Superiority; p < 0.05, Regression, Logistic

5. Other Pre Specified Outcome: Change in Depressive Symptoms
Description: Participants self-reported level of depressive symptoms at pre-test and post-test using the brief version of the Mood and Feelings Questionnaire (b-MFQ; Angold et al., 1995). The measure include 13 items on a scale of 0 to 2, with a total range of 0 to 26. Scores of 12 or greater suggest clinical depression, so higher scores indicate higher depressive symptoms, which is a negative outcome.
Time Frame: Collected at Pre-Test and Post-Test visits (within approximately 1 month of active treatment).
Population: N = number of students who completed the survey. We are missing 1 survey from an intervention participant at post-test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
Number analyzed (Participants) | 23 | 48
score on a scale
  Pre-test | 4.7 (4.1) | 5.7 (4.1)
  Post-test: number analyzed (Participants) | 23 | 47
  Post-test | 4.0 (3.0) | 5.3 (4.0)
Statistical Analysis 1: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; Test type: Superiority; p = 0.70, ANOVA — Group by time interaction; Repeated measures ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at the beginning of the study start date until the last follow-up employment data was collected, an average of 12 months.
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/48
Other Adverse Events (participants affected / at risk) | 0/23 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03514134/Prot_SAP_000.pdf
  • Informed Consent Form: Student Consent Form (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT03514134/ICF_001.pdf
  • Informed Consent Form: Student Assent Form (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT03514134/ICF_002.pdf